CLINICAL TRIAL: NCT03098511
Title: CT-Perfusion for Neurological Diagnostic Evaluation: a Prospective Canadian Multicenter Diagnostic Test Study
Brief Title: CT-Perfusion for Neurological Diagnostic Evaluation
Acronym: INDex-CTP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 16.379
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Neurological Determination of Death
Keywords: Neurological Determination of Death; Determination of Death; CT-Perfusion scan; Ancillary Test; Organ Donation
MeSH Terms: conditions — Death

STUDY DESIGN:
Masking Description: 1. Participant will be comatose
  2. Care providers, investigators and outcome assessors will be blinded from the results of the CT-Perfusion scan result (for the clinical assessment) and from the clinical assessment results (for the CT-Perfusion scan interpretation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurological Diagnostic Evaluation (Other): Exams performed according to a determined schedule following admission in the intensive care unit in order to validate CT-perfusion as an accurate ancillary test for neurological diagnostic.
  Interventions: Diagnostic Test: Neurological Diagnostic Evaluation

INTERVENTIONS:
Diagnostic Test: Neurological Diagnostic Evaluation — Clinical Data:
  * Demographic data
  * Daily data (clinical exams, laboratory data)
  * Drug administration
  * Additional clinical or ancillary neurological determination test
  Diagnostic Intervention:
  * CT-Perfusion
  * CT-Angiography reconstructions
  Reference Standard:
  - Clinical Neurological Exam
  Blood Samples (Pharmacokinetics, Inflammatory & Nanovesicles Parameters):
  * At the time of patient enrolment
  * 6 hours after patient enrolment
  * At the time of the clinical neurological exam
  Secondary Outcome measures at 6 months:
  * extended Glasgow Outcome Scale (GOSe)
  * modified Rankin Scale (mRS)

SUMMARY:
For the purpose of organ donation after neurological determination of death (NDD), death must be declared using a set of standardized clinical criteria. When a full clinical evaluation cannot be completed, additional neuroimaging ancillary testing is required. The ideal ancillary test for NDD would demonstrate no cerebral blood flow, be free of false-positive and false negative results, rapid, safe, readily available, non-invasive, and inexpensive. No current ancillary test for NDD meets these criteria. Computed tomography (CT) perfusion has the characteristics of an ideal test for NDD, but has not been evaluated for routine clinical use for NDD.

The overarching goal of this project is to improve the NDD process by establishing CT-perfusion as the ideal ancillary test. A large prospective Canadian multi-centre diagnostic cohort study will be conducted to validate CT-perfusion for the neurological determination of death.

Specific objectives are:

Primary objective: To determine diagnostic accuracy of CT-perfusion compared to complete clinical evaluation for NDD.

Secondary objectives: 1) To confirm the safety of performing CT-perfusion in critically ill patients suspected of being neurologically deceased; 2) To establish the CT-perfusion inter-rater reliability for NDD; 3) To evaluate the diagnostic accuracy of CT-angiography compared to complete clinical evaluation and to CT-perfusion for NDD; 4) To describe the clearance of commonly used sedatives and narcotics in the setting of NDD; and 5) to investigate biological changes (inflammatory and nanovesicles) that occur in humans during the brain dying process.

DETAILED DESCRIPTION:
The investigators will conduct a large prospective Canadian multi-centre diagnostic cohort study. The primary diagnostic test evaluated will be CT-perfusion. The reference standard will be the complete clinical evaluation of brainstem functions. Comatose patients at high risk of neurological death exempt of confounding factors (e.g. hypothermic patients, use of long-acting sedatives, etc.) will be included. All patients will undergo CT-perfusion of the head (with CT-angiography reconstructions) followed by a complete NDD assessment. Both CT-perfusion and the clinical exam will be performed by independent assessors blinded from each others' interpretation. The primary endpoints will be the sensitivity and specificity of CT-perfusion to confirm NDD. Safety endpoints will be CT-perfusion -related adverse events (i.e. contrast-induced kidney injury, new hemodynamic instability while undergoing CT-perfusion). The true negative, true positive, false negative and false positive for CT-angiography obtained from the CT-perfusion source images when compared to the reference standard as well as when compared to the CT-Perfusion will also be reported. The sensitivity and specificity of CT-angiography compared to the reference standard and to CT-perfusion along with corresponding 95% confidence intervals will be calculated. Individual patient and population pharmacokinetics of analgesics and sedatives will be determined. To better investigate the impact of residual circulating sedative or narcotic levels on the accuracy of CT-Perfusion and CT-Angiography, Receiver Operating Characteristics (ROC) curves for varying levels of narcotic or sedative thresholds and compute the ROC area under the curve for each threshold will be plotted. To assess the immune phenotype, peripheral blood mononuclear cells activation will be evaluated by flow cytometry and cytokines by multiplex analyses. Nanovesicles fraction will be isolated from the plasma by ultracentrifugation and antigenic content and enzymatic activity. The plasma will finally be analysed by ELISAs and multiplex analyses to determine the levels of pro-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years and older
2. Admitted in the intensive care unit with a brain injury
3. Glasgow Coma Scale (GCS) = 3
4. Sedation stopped for at least 6 hours

Exclusion Criteria:

1. Patients with the following contraindications to CT-perfusion will be excluded from the study:

   * Pregnancy
   * Contrast allergy
   * Clinician refuses inclusion because of kidney injury.
2. Patients with any of the following confounding factors precluding complete clinical neurological evaluation will be excluded from the study:

   * Cervical fracture above C6
   * Significant facial trauma limiting cranial nerve examination
   * Hypothermia < 34 °C
   * Use of intravenous barbiturates at any time since admission
   * Unresuscitated shock
   * Peripheral nerve or muscle dysfunction or neuromuscular blockade potentially accounting for unresponsiveness
   * Anoxic brain injury < 24h (or 72h if therapeutic hypothermia)
   * Attending physician disagrees to conduct an apnea test
   * Any other abnormalities deemed a confounding factor for NDD by the attending clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CT-perfusion | CT-Perfusion scan and clinical assessment must be less than 2 hours apart
  Sensitivity and specificity for brainstem death of CT-perfusion compared to the clinical examination

SECONDARY OUTCOMES:
Predictive Values | CT-Perfusion scan and clinical assessment must be less than 2 hours apart
  Positive and negative predictive values between two independent neuroradiology interpretations of CT-perfusion for brainstem death
Likelihood Ratios | CT-Perfusion scan and clinical assessment must be less than 2 hours apart
  Positive and negative likelihood ratios between two independent neuroradiology interpretations of CT-perfusion for brainstem death
Inter-rater Agreement | CT-Perfusion scan and clinical assessment must be less than 2 hours apart
  Between two independent neuroradiology interpretations of CT-perfusion for brainstem death
Volume of Distribution | 48 hours
  Volume of distribution from serum concentrations and drug dosing history
Clearance | 48 hours
  Volume of plasma completely cleared of the drug expressed as mL/min
Elimination Rate Constant | 48 hours
  Rate at which the drug is removed from the body
Concentration-time Curve | 48 hours
  Concentration of drug versus time
Accuracy of CT-perfusion at 6 Months | 6 months
  Sensitivity and specificity for brainstem death of CT-perfusion compared to the clinical examination for a good mRS score (3 or less) at 6 months
Accuracy of the Predictive Values at 6 Months | 6 months
  Positive and negative predictive values between two independent neuroradiology interpretations of CT-perfusion for brainstem death for a good mRS score (3 or less) at 6 months
Accuracy of the Likelihood Ratios at 6 Months | 6 months
  Positive and negative likelihood ratios between two independent neuroradiology interpretations of CT-perfusion for brainstem death for a good mRS score (3 or less) at 6 months
Accuracy of the Inter-rater Agreement at 6 Months | 6 months
  Between two independent neuroradiology interpretations of CT-perfusion for brainstem death for a good mRS score (3 or less) at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaël Chassé, MD PhD FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Jai JS Shankar, MD MSc FRCPC, Principal Investigator — University of Manitoba
Locations (14):
- Canada (14):
  - Foothills Medical Centre, Calgary, Alberta
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Health System, Brampton, Ontario
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St-Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No